CLINICAL TRIAL: NCT07012681
Title: Investigation of the Effects of Discharge Education Strategies on Quality of Life and Daily Living Activities in Patients Who Have Undergone Intracranial Surgery. This Study Was Designed as a Randomized Controlled Trial to Determine the Most Effective Method Verbal Education or a Combination of Verbal Education and Written Brochure Educationon the Quality of Life and Daily Living Activities of Patients Who Have Undergone Intracranial Surgery
Brief Title: Investigation of the Effects of Discharge Education Strategies on Quality of Life and Daily Living Activities in Patients Who Have Undergone Intracranial Surgery.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Working hours have been shortened due to various reasons
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Hanife Damla Çaygör, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Caygor/08.05.2025
Record Dates: First submitted 2025-05-13; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Surgery
Keywords: Patient discharge management
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Arm 1: Oral Training Group Arm 2: Oral and Written Brochure training Group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- discharge education (oral education) (Experimental): oral training group
  Interventions: Other: discharge education (oral education)
- discharge training (oral and written training) (Experimental): The group that received oral and written brochure training
  Interventions: Other: discharge training (oral and written brochure)

INTERVENTIONS:
Other: discharge training (oral and written brochure) — The group that received oral and written brochure training during discharge training
  Arms: discharge training (oral and written training)
Other: discharge education (oral education) — group receiving oral training in discharge training
  Arms: discharge education (oral education)

SUMMARY:
It was planned to provide education using verbal education or verbal and picture-text brochure method as a discharge education strategy for patients who underwent intracranial surgery. In this context, it was aimed to compare the effects of two discharge education strategies used in the discharge education of patients who underwent intracranial surgery on the quality of life and daily living activities of the patients.

DETAILED DESCRIPTION:
In this study, it was planned to provide education to patients who underwent intracranial surgery by using verbal education or verbal and pictorial brochure methods as a discharge education strategy. The evaluation of the effect of this education, which includes content on skin wound care, nutrition, drainage, exercise, medication management and seizures, on the quality of life and daily living activities of the patients In this context, it was aimed to compare the effects of two discharge education strategies used in the discharge education of patients who underwent intracranial surgery on the quality of life and daily living activities of the patients.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

* Have undergone intracranial surgery
* Voluntarily agree to participate in the study
* Be between 18 and 75 years of age
* Be literate and speak Turkish
* Be open to communication and cooperation
* Be mentally healthy
* Have no visual, hearing, or speech impairments

Exclusion Criteria

Participants will be excluded from the study if they meet any of the following:

* Refuse to participate in the study
* Are not native Turkish speakers
* Are illiterate
* Have visual, hearing, or speech impairments
* Have a diagnosed psychological disorder
* Have been diagnosed with dementia or Alzheimer's disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
quality of life scale and activities of daily living scale | Assessed for 1 month after hospital discharge
  There are (0-100) points on the quality of life scale, and as the score increases, the quality of life increases. There are (0-6) points on the daily living activities scale, and as the score increases, the functionality increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Eğitim ve Araştırma Hastanesi, Istanbul, Sultangazi, Turkey (Türkiye)